CLINICAL TRIAL: NCT06761755
Title: Combined Effects of Kinesiology Taping and Progressive Muscle Relaxation Technique on Pain, Anxiety and Body Awareness in Primary Dysmenorrhea
Brief Title: Taping and PMR Effects in Primary Dysmenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/khushbu sohail
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Dysmenorrhea Primary
Keywords: : Anxiety, dysmenorrhea, pain,
MeSH Terms: conditions — Anxiety Disorders; Dysmenorrhea; Pain | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Hot pack+ kinesiology taping + progressive muscle relaxation technique Group A has given the kinesiology taping on the lower abdomen and back for 1-3 days with progressive muscle relaxation technique for 10-20 minutes and a baseline treatment hot pack at a time twice a day from the start of menstruation
  Interventions: Other: hot pack , K taping , Progressive muscle relaxation
- Group B (Experimental): hot pack + kinesiology taping Group B has receive the kinesiology taping on the lower abdomen and baseline treatment hot pack without progressive muscle relaxation technique for 1-3 days
  Interventions: Other: hot pack , K taping , Progressive muscle relaxation

INTERVENTIONS:
Other: hot pack , K taping , Progressive muscle relaxation — Group A has given the kinesiology taping on the lower abdomen and back for 1-3 days with progressive muscle relaxation technique for 10-20 minutes and a baseline treatment hot pack at a time twice a day from the start of menstruation
  Group B has receive the kinesiology taping on the lower abdomen and baseline treatment hot pack without progressive muscle relaxation technique for 1-3 days

SUMMARY:
The study is randomized controlled trial,The study conducted in two groups. Group A has given the kinesiology taping on the lower abdomen and back for 1-3 days with progressive muscle relaxation technique for 10-20 minutes and a baseline treatment hot pack at a time twice a day from the start of menstruation and Group B has receive the kinesiology taping on the lower abdomen and baseline treatment hot pack without progressive muscle relaxation technique for 1-3 days. The total treatment duration will be 6 weeks. The rationale of this study is to provide empirical evidence regarding the efficacy and safety of kinesiology taping and progressive muscle relaxation. By investigating the potential benefits of this intervention, healthcare professionals can make informed decisions about incorporating K-taping and PMR in primary dysmenorhea. Focusing on the impact of kinesiology taping and progressive muscle relaxation on pain,anxiety, and body awareness aligns with a patient-centered approach to care. The goal is not only to reduce symptoms but also to enhance overall well-being and functional capacity

DETAILED DESCRIPTION:
The literature gap of the study is that upto our knowledge, there is little or no evidence found in previous researches on the combined effects of kinesiology taping in combination with progressive muscle relaxation technique in primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* • Aged between 18-25 years

  * Unmarried female
  * Taking ≥4 points from Visual Analog Scale during menstrual cycle
  * Had moderate menstrual pain as measured by WaLLID score

Exclusion Criteria:

* • Complaints of low back pain due to any other pathology, any skin infection, sensitive skin or allergic to Kinesio Tape.

  * PCOD, Uterine/ ovarian tumor, Acute/ chronic pelvic pathology like PID, endometriosis, spinal pathology and deformity
  * Endometrial polyp, having a pelvic infection, using an intrauterine device, having venous congestion in the internal genital organs.
  * Who take analgesic

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females with primary dysmenorrhea
Enrollment: 30 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
numerical pain rating scale | 1st day
  changes from base line NPRS is used to access the pain at 1st day or before the start of menstruation at the end score is calculated by dividing the obtained score by total 0 means no pain and 10 is maximum
STAI tool (state triate anxiety inventory) | 1st day
  changes in the baseline ,STAI tool to access the anxiety of the patient feels at the start of menstruation at the end the score is calculated by dividing the score by total 0 means no anxiety and 4 means maximum anxiety
Body awareness questionaire | 1st day
  Changes in the baseline, Body Awareness Questionnaire (Shields, Mallory & Simon, 1989) acess the body awarenss during dysmenorhea , at the end the score is calcuted 0 means not true of me and 7 is the maximum true of me

SECONDARY OUTCOMES:
Wallid questionaire | 1st day
  walid to access the Working ability, Location, Intensity (Wong-Baker) and Days of pain Score: 0 without dysmenorrhea, 1-4 mild dysmenorrhea, 5-7 moderate dysmenorrhea, 8-12 severe dysmenorrhea. Wong-Baker scale was reclassified to adjust a four-level scale.

CONTACTS AND LOCATIONS:
Overall Officials: Iqra Abdul ghafoor, PPDPT, Principal Investigator — Riphah International University
Locations (1):
- Ghurki hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pazare S, Sawant L, Ingale S. The Effects of Kinesio Taping and Isometric Exercises on Pain in Primary Dysmenorrhea-A Comparative Study. Website: www ijpot com. 2019;13(4):4117
- [Background] Bandara EMIA, Kularathne WNI, Brain K, Weerasekara I. Safety and efficacy of therapeutic taping in primary dysmenorrhea: a systematic review and meta-analysis. Sci Rep. 2022 May 3;12(1):7146. doi: 10.1038/s41598-022-11034-w. PMID 35504906
- [Background] Dogan H, Eroglu S, Akbayrak T. The effect of kinesio taping and lifestyle changes on pain, body awareness and quality of life in primary dysmenorrhea. Complement Ther Clin Pract. 2020 May;39:101120. doi: 10.1016/j.ctcp.2020.101120. Epub 2020 Feb 22. PMID 32379659
- [Background] Mejias-Gil E, Garrido-Ardila EM, Montanero-Fernandez J, Jimenez-Palomares M, Rodriguez-Mansilla J, Gonzalez Lopez-Arza MV. Kinesio Taping vs. Auricular Acupressure for the Personalised Treatment of Primary Dysmenorrhoea: A Pilot Randomized Controlled Trial. J Pers Med. 2021 Aug 19;11(8):809. doi: 10.3390/jpm11080809. PMID 34442453
- [Background] Ferries-Rowe E, Corey E, Archer JS. Primary Dysmenorrhea: Diagnosis and Therapy. Obstet Gynecol. 2020 Nov;136(5):1047-1058. doi: 10.1097/AOG.0000000000004096. PMID 33030880
- [Background] Toprak Celenay S, Kavalci B, Karakus A, Alkan A. Effects of kinesio tape application on pain, anxiety, and menstrual complaints in women with primary dysmenorrhea: A randomized sham-controlled trial. Complement Ther Clin Pract. 2020 May;39:101148. doi: 10.1016/j.ctcp.2020.101148. Epub 2020 Mar 18. PMID 32379680
- [Background] Hamdy Nasr Abdelhalim E, Yehia Moustafa Sweelam M, Abd Elaziem Mohamed A, Gomaa Mohamed Amer F, El-Shabory ME-S, El-Hoda N. Effect of Progressive Muscle Relaxation Technique on Pain Intensity and FatigueAssociated with Primary Dysmenorrhea among Female Adolescents. Egyptian Journal of Health Care. 2023;14(1):486-500
- [Background] Guruprasad P, Sharma U, Palekar T, Pimpri P. Immediate Effect of Yoga Postures v/s Physiotherapy Exercises Along with K-Taping on Pain in Dysmenorrhea. International Journal of Scientific Research in Science and Technology. 2019;6(2):487-94.
- [Background] Unal A, Altug F, Erden A, Cavlak U, Senol H. Validity and reliability of the Body Awareness Questionnaire in patients with non-specific chronic low back pain. Acta Neurol Belg. 2021 Jun;121(3):701-705. doi: 10.1007/s13760-020-01399-y. Epub 2020 Jun 21. PMID 32566989
- [Background] Patel R, Patel AK, Gupta K. Premenstrual symptoms and general health among young adolescent girls: A correlational study. Perspectives on Coping Strategies for Menstrual and Premenstrual Distress: IGI Global; 2023. p. 1-12.
- [Background] Sakpal S, Patil C. Efficacy of Chair Aerobics and Progressive Muscle Relaxation in Primary Dysmenorrhea. Journal of Coastal Life Medicine. 2023;11:1511-6.
- [Background] George SA, Suresh G, Fathima P, Alias H. Effectiveness of physical activity and relaxation techniques in primary dysmenorrhea among college students. Int J Sci Res. 2019;8(11):531-3.
- [Background] Kaur A, Ray G, Mitra M. Comparing the effectiveness of connective tissue mobilisation and kinesio-taping on females with primary dysmenorrhea. Indian Journal of Physiotherapy & Occupational Therapy. 2017;11:70-5
- [Background] Temizkan S, BUDAK M. The Effects of Kinesiological Taping and Aerobic Exercise in Women with Primary Dysmenorrhea: A Randomized Single-Blind Controlled Trial. 2021.
- [Background] Yildiz E, Acaroglu R. The Effect of Massage and Progressive Relaxation Exercises on Pain Intensity and Menstrual Symptoms in Students With Primary Dysmenorrhea: A Randomized Controlled Trial. Holist Nurs Pract. 2022 Sep-Oct 01;36(5):284-294. doi: 10.1097/HNP.0000000000000541. PMID 35981113
- [Background] Jiang J, Zhuang Y, Si S, Cheng H, Alifu X, Mo M, Zhou H, Liu H, Yu Y. The Association of Reproductive Hormones During the Menstrual Period with Primary Dysmenorrhea. Int J Womens Health. 2023 Oct 9;15:1501-1514. doi: 10.2147/IJWH.S421950. eCollection 2023. PMID 37840555
- [Background] Ibrahim ZM, Alharkan BS, Alanzi EH, Alnasban HA, Alsuwailem MM, Al Khalil WK. Efficacy of active stretching exercises against symptoms of primary dysmenorrhoea in young adult females: a randomized controlled trial. Physiotherapy Quarterly. 2023;31(3).
- [Background] Kirca N, Celik AS. The effect of yoga on pain level in primary dysmenorrhea. Health Care Women Int. 2023 May;44(5):601-620. doi: 10.1080/07399332.2021.1958818. Epub 2021 Sep 17. PMID 34534030
- [Background] Aldinda TW, Sumarni S, Mulyantoro DK, Azam M. Progressive muscle relaxation application (PURE App) for dysmenorrhea. 2022.
- [Background] Kustriyanti D, Boediarsih B. Muscle Relaxation Therapy for Dysmenorrhea. Health Notions. 2017;1(4):315-20
- [Background] Celik AS, Apay SE. Effect of progressive relaxation exercises on primary dysmenorrhea in Turkish students: A randomized prospective controlled trial. Complement Ther Clin Pract. 2021 Feb;42:101280. doi: 10.1016/j.ctcp.2020.101280. Epub 2020 Nov 30. PMID 33310052
- [Background] Arshad S, Qureshi MF, Deeba F, Sarshad S, Shiraz S, Farooq S, et al. To compare the effectiveness of taping technique and hydrotherapy in treatment of primary dysmenorrhea. Inter J Endor Health Sci Res. 2018;6(3):34-42.
- [Background] Kumar S, Kanti V, Potturi G, Kumar P. Effect of Kinesio tape application on quality of life and functional independence among Nulligravida women with Primary dysmenorrhea: A randomized control trial. Journal of Disability Studies. 2023;9(1):13-6